CLINICAL TRIAL: NCT06543615
Title: Preoperative Ultrasound Evaluation of Fasting Residual Gastric Volume in Patients With Previous Sleeve Gastrectomy : Comparative Study With Patients Without History of Bariatric Surgeries
Brief Title: Preoperative Ultrasound Evaluation of Fasting Residual Gastric Volume in Patients With Previous Sleeve Gastrectomy
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: Fasting required preoperative
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-11

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Patients undergoing laparoscopic cholecystectomy with history of sleeve gastrectomy: Gastric residual volume will be assessed after 8 hours of fasting preoperatively using ultrasonography in patients undergoing laparoscopic cholecystectomy with history of sleeve gastrectomy
  Interventions: Device: Ultrasonography
- Patients undergoing laparoscopic cholecystectomy with no history of bariatric surgeries: Gastric residual volume will be assessed after 8 hours of fasting preoperatively using ultrasonography in patients undergoing laparoscopic cholecystectomy with No history of bariatric surgeries
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Ultrasound assessment of residual gastric volume

SUMMARY:
Preoperative US assessment of residual gastric volume in both; patients with previous laparoscopic sleeve gastrectomy and those without history of bariatric surgeries, undergoing elective laparoscopic cholecystectomy, aiming to develop a step for recommendations for fasting guidelines

DETAILED DESCRIPTION:
No doubt, that perioperative aspiration of gastric content during anesthesia process is every anesthesiologist's nightmare, which can lead to serious morbidities and mortalities with a rate of 5% to 9 % in anesthesia airway management accidents.

Risk of aspiration usually present during induction of anesthesia due to passive regurgitation during endotracheal intubation while it may occur during recovery from anesthesia in patients with active vomiting.

It is known that the volume of residual gastric content is one of the most important factors that can lead to significant increase in the risk of perioperative pulmonary aspiration, acknowledging this fact, lead the American society of Anesthesiology (ASA) to recommend for eight hours fasting for solids (fats and/or meats), six hours for non-human milk and light meals, and two hours for clear fluids, to reduce residual gastric volume and subsequently the risk of perioperative aspiration.

There are many different ways to asses gastric content for example nasogastric tube aspiration of gastric content which is an invasive technique. Other ways include imaging tools like abdominal CT scan which is not easily done and will have extra cost on the patient . In addition, wireless motility capsules and gastric emptying scintigraphy can be used but all of them are not suitable for routine assessment.

On the other hand Point-of-Care (POC) ultrasound usage in anesthesia management has provided a wide range of rapid, bed side and non-invasive, easy and fast techniques that help to reduce the risk of morbidity and mortality. It also, helped to provide a technique for qualitative and quantitative assessments of residual gastric contents preoperatively through gastric antrum US assessment using measurement of the antral cross-sectional area.

In the past it was believed that gastric content more than 2.5 ml/kg was considered as an "at risk" stomach volume , but nowadays several studies using ultrasonography assessment of residual gastric content indicated that the accepted volume should be less than 1.5 ml/kg in healthy fasting adult to define an empty stomach.

It is well known that bariatric surgeries nowadays became very popular among patients suffering from obesity for the sake of better quality of life specially sleeve gastrectomy and Roux-en-Y gastric bypass surgeries. A statistical study was done among the American population in 2018 reported that about 252 000 bariatric procedures are being performed every year and the number is rising by time specially with advanced surgical techniques that reduced the complications of these types of surgeries. However; no statistics has been released for Egyptian population.

As regards, Nele, et. al. reported that gastric emptying was significantly reduced in patients with history of sleeve gastrectomy and Roux-en-Y gastric bypass surgeries as compared to obese patients by comparing gastric emptying scintigraphy, wireless motility capsule and gastrointestinal fluid aspiration techniques.

Also Eric, et al. in their meta-analysis study, have reported that gastric emptying time was reduced after gastric bypass surgery but it was constant or increased with endoscopically inserted intragastric balloons.

Many studies tried to asses changes in GIT physiology after bariatric surgeries including gastric emptying time using several methods as mentioned before but less frequently ultrasound guided assessment.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists physical status classification) I-II
* Aged between 21 and 45 years old undergoing elective surgery.
* Fasting 8 hours preoperative.
* Body mass index less than 35 Kg/m2

Exclusion Criteria:

* ASA physical status more than II .
* Pregnant women.
* Patients above 45 years and below 21 years.
* History of drug intake of prokinetics or any drug that affect gastric emptying and/or motility.
* Diabetic patients.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups both undergoing laparoscopic cholecystectomy the first group with history of laparoscopic sleeve gastrectomy, while the second group with No history of previous bariatric surgeries according to inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
residual gastric volume | After fasting 8 hours immediately preoperative
  Measurement of residual gastric volume immediately preoperative in right lateral decubitus after fasting 8 hours

SECONDARY OUTCOMES:
incidence of aspiration | Perioperative ( immediately preoperative, intraoperative or during recovery from anesthesia post operative
  Documentation of aspiration incidence immediately preoperative, intraoperative or during recovery from anesthesia post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma G, Jacob R, Mahankali S, Ravindra MN. Preoperative assessment of gastric contents and volume using bedside ultrasound in adult patients: A prospective, observational, correlation study. Indian J Anaesth. 2018 Oct;62(10):753-758. doi: 10.4103/ija.IJA_147_18. PMID 30443057
- [Background] Walter U, Loong C, Loewenhaupt M, Schlabitz W. Evidence of a magnetic gaplike excitation in URu2Si2. Phys Rev B Condens Matter. 1986 Jun 1;33(11):7875-7878. doi: 10.1103/physrevb.33.7875. No abstract available. PMID 9938176
- [Background] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530
- [Background] Steenackers N, Vanuytsel T, Augustijns P, Deleus E, Deckers W, Deroose CM, Falony G, Lannoo M, Mertens A, Mols R, Vangoitsenhoven R, Wauters L, Van der Schueren B, Matthys C. Effect of sleeve gastrectomy and Roux-en-Y gastric bypass on gastrointestinal physiology. Eur J Pharm Biopharm. 2023 Feb;183:92-101. doi: 10.1016/j.ejpb.2022.12.018. Epub 2023 Jan 2. PMID 36603693